CLINICAL TRIAL: NCT01089036
Title: Oxidant-antioxidant Activity, Free Radicle Activity, Immune Response and Biomarkers in ECMO Patients
Brief Title: Oxidant-antioxidant Activity, Free Radicle Activity, Immune Response and Biomarkers in Extracorporeal Membrane Oxygenation (ECMO) Patients
Acronym: ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200911043R
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction; Myocarditis; Cardiomyopathy
Keywords: ECMO; cardiogenic shock; ROS; GPx; cytokines
MeSH Terms: conditions — Shock, Cardiogenic; Myocarditis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,plasma, and cells for study. Once the study is completed, biospecimen will be discarded.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- survival: ECMO survival patients
- ECMO non-survival: ECMO non-survivals

SUMMARY:
We would like to investigate novel diagnostic methods or biomarkers to early predict the success of ECMO therapy for cardiogenic shock patients during the early stage after ECMO treatment.

DETAILED DESCRIPTION:
In the investigators previous study (Ann Thorac Surg 2002, 73: 538-545), the investigators knew that for those adult patients receiving ECMO support for post-cardiotomy cardiogenic shock, 1/3 of them would survive to discharge, 1/3 could not be weaned from ECMO and died on the ECMO support, and 1/3 could be weaned from ECMO support, but finally died of multiple organ failure. However, by clinical observation in the first few days of ECMO support, it would be very difficult to predict the outcome of a specified individual patient. Therefore, the investigators usually wait for four to six days to know whether the ECMO treatment is successful or not. If the investigators could predict the result one or two days earlier, this would give physicians enough time to make medical decision. Therefore, the early parameters that could be used to predict the outcome of ECMO treatment would be very valuable. The investigators also found that despite obscure clinical presentation, there was a significant difference in serum cytokines' concentration on the 3rd day of ECMO support between "ECMO successful" and "ECMO failure" patients.

In this study, the investigators will further investigate leukocyte free radical activity, oxidation damage marker (8-OHdG concentration) in serum, whole blood glutathione peroxidase activity for antioxidation, serum IL-6, IL-12, IL-8, IL-10, transforming growth factor-β and other biochemical concentrations and immune cellular changes during the period of ECMO treatment. Patient's blood samples before and 2, 6, 12, 24, 48, 72 hours after ECMO support treatment, at ECMO removal and ICU discharge will be collected and used for the study. The measured factors and the final outcome will be compared. The investigators hope to find early factors change during ECMO treatment among biochemical, immunological and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≧ 18 yr. 2. cardiogenic shock, needing ECMO support

Exclusion Criteria:

* 1. pre-existing sepsis 2. pre-existing chronic renal failure (dialysis dependent), liver failure, multiple organ failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  1. ≧ 18 yr.
  2. cardiogenic shock, needing ECMO support
  Exclusion criteria
  1. pre-existing sepsis
  2. pre-existing chronic renal failure (dialysis dependent), liver failure, multiple organ failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mortality or multi-organ failure | 7 days
  Patients who survived for more than 7 days after ECMO treatment were defined as survival, and non-survival patients were defined as expired or multiple organ failure incompatible with life within 7 days after ECMO installation.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Je Ko, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan